CLINICAL TRIAL: NCT01271504
Title: An Open-Label, Multicenter, Randomized, Phase Ib/II Study of E7050 in Combination With Sorafenib Versus Sorafenib Alone as First Line Therapy in Patients With Hepatocellular Carcinoma
Brief Title: E7050 in Combination With Sorafenib Versus Sorafenib Alone as First Line Therapy in Participants With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: PharmaBio Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7050-701; 2011-000752-41 (EudraCT Number)
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2017-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Cancer; liver; hepatocellular carcinoma; phase I; phase II
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase Ib: Cohort 1,2, and 3 (Active Comparator): Phase Ib: Cohort 1; 200 mg E7050 + 400 mg Sorafenib Cohort 2; 300 mg E7050 + 400 mg Sorafenib Cohort 3; 400 mg E7050 + Sorafenib
  Interventions: Drug: Sorafenib
- Phase II: Arm 1; E7050 + Sorafenib (Active Comparator): Phase II: Arm 1; E7050 + 400 mg Sorafenib Arm 2; 400 mg Sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Phase Ib: Cohort 1; 200 mg E7050 + 400 mg Sorafenib Cohort 2; 300 mg E7050 + 400 mg Sorafenib Cohort 3; 400 mg E7050 + Sorafenib
  Arms: Phase Ib: Cohort 1,2, and 3
Drug: Sorafenib — E7050 given orally at 200, 300 or 400 mg once daily.
  Sorafenib given orally, 400 mg twice daily.
  Arms: Phase II: Arm 1; E7050 + Sorafenib

SUMMARY:
The purpose of this study is to determine whether patients with hepatocellular carcinoma who receive either E7050 administered with Sorafenib or Sorafenib alone experience greater benefit (cancer responds to treatment) when E7050 is administered with Sorafenib.

DETAILED DESCRIPTION:
This open-label, multicenter, randomized study will consist of a Phase Ib: a safety run-in period with 3 ascending doses of E7050 in combination with sorafenib; and a Phase II portion: a randomized 2-arm period. Approximately 95 patients with hepatocellular carcinoma will be enrolled in the study (10-15 patients in the Phase Ib portion and 80 patients in the Phase II portion). Patients will only participate in either the Phase Ib or the Phase II portion of the study. In both Phase Ib and phase II, Patients will receive study treatment (E7050 plus sorafenib or sorafenib alone) until the occurrence of progressive disease (PD)for approximately six 28-day cycles (24 weeks). After 6 cycles. ath the discretion of the Investigator and in consultation with the Medical Monitor, patients who are experiencing clinical benefit may continue E7050, with or without sorafenib (Arm 1), or may continue sorafenib alone (Arm 2), depending on the original randomization treatment arm, for as long as clinical benefit is sustained and the treatment is well tolerated. Patients will be followed until death following completion of therapy.

ELIGIBILITY:
Inclusion Criteria

* Unresectable locally advanced or metastatic HCC;
* Histologic confirmation not required if other diagnostic criteria are met;
* No previous systemic anti-cancer therapy permitted (2 prior systemic anti-cancer regimen are allowed in Phase Ib). Previous chemoembolization, radioembolization, radiofrequency ablation, or other local ablative therapies are permitted if greater than 6 weeks of first day of study-defined treatment;
* ECOG PS 0 or 1; Child-Pugh Cirrhotic Status A or B with a score of 7;
* Blood pressure must be well-controlled (less than or equal to 140/90 mmHg at screening) with or without antihypertensive medication. Patients must have no history of hypertensive crisis or hypertensive encephalopathy;

Exclusion Criteria

* Previously received E7050 anti-cmet, or anti-angiogenic therapy (prior anti-angiogenic therapy is permitted in Phase Ib only);
* Presence of brain metastases, unless the patient has received adequate treatment at least 4 weeks prior to randomization, and is stable, asymptomatic, and off steroids for at least 4 weeks prior to randomization;
* Palliative radiotherapy is not permitted throughout the study period;
* Active hemoptysis
* Serious non-healing wound, ulcer, or active bone fracture;
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to commencing study treatment, or anticipation of need for a major surgical procedure during the course of the study;
* Clinically significant gastrointestinal bleeding (bleeding requiring procedural intervention, eg. variceal banding, transjugular intrahepatic portosystemic shunt (TIPS) procedure, arterial embolization, topical coagulation therapy) within 6 months prior to first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-07-19 (Actual); Primary Completion 2015-06-23 (Actual); Study Completion 2015-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Versola, RN, Study Director — Quintiles, Inc.
Locations (20):
- United States (7):
  - Tucson, Arizona
  - Fort Myers, Florida
  - St. Petersburg, Florida
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Nashville, Tennessee
- Belgium (2):
  - Brussels
  - Leuven
- Italy (3):
  - Rozzano, Milano
  - Modena
  - Pavia
- Madrid, Spain
- Ukraine (4):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Lviv
- United Kingdom (3):
  - London, Greater London
  - Manchester, Greater Manchester
  - Glasgow, Strathclyde

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in Belgium, Italy, Spain, the Ukraine, the United Kingdom and the United States from 19 July 2011 to 23 June 2015.
Pre-assignment Details: A total of 102 participants were enrolled and randomized in this study, out of which, 15 participants were enrolled in Phase 1b of study, of which 14 received study drug, and 87 participants were enrolled in Phase 2 of study, of which 84 participants received the study drug.
Groups:
- Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg: Participants received golvatinib 200 milligram (mg), tablet, orally, once daily in combination with sorafenib 400 mg, tablet, orally, twice daily in 28-days treatment cycles until the occurrence of progressive disease (PD), unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first (Up to 513 Days).
- Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg: Participants received golvatinib 300 mg, tablet, orally, once daily in combination with sorafenib 400 mg, tablet, orally, twice daily in 28-days treatment cycles until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first (Up to 513 Days).
- Phase 2: Golvatinib 200 mg + Sorafenib 400 mg: Participants received golvatinib 200 mg, tablet, orally, once daily in combination with sorafenib 400 mg, tablet, orally, twice daily in 28-days treatment cycles until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first (Up to 705 Days).
- Phase 2: Sorafenib 400 mg: Participants received sorafenib 400 mg, tablet, orally, twice daily in 28-days treatment cycles until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first (Up to 705 Days).
Period: Overall Study
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Started | 7 | 8 | 44 | 43
Treated | 7 | 7 | 42 | 42
Completed | 0 | 0 | 0 | 0
Not Completed | 7 | 8 | 44 | 43
Not completed — Death | 7 | 6 | 32 | 32
Not completed — Lost to Follow-up | 0 | 1 | 3 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Administrative Reasons | 0 | 0 | 6 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3
Not completed — Other | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants enrolled and randomized into the Phase 1b and Phase 2 of this study, except those who dropped out of the study prior to receiving any study drug, or were without any safety assessment after first dose of study drug.
Groups:
- Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg: Participants received golvatinib 200 mg, tablet, orally, once daily in combination with sorafenib 400 mg, tablet, orally, twice daily in 28-days treatment cycles until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first (Up to 513 Days).
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg | Total
Number analyzed (Participants) | 7 | 7 | 42 | 42 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (15.68) | 68.1 (9.56) | 63.2 (9.31) | 65.8 (8.02) | 63.9 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 10 | 12 | 25
  Male | 6 | 5 | 32 | 30 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 5 | 8
  Not Hispanic or Latino | 7 | 5 | 36 | 36 | 84
  Unknown or Not Reported | 0 | 0 | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 4 | 1 | 5
  White | 7 | 5 | 37 | 37 | 86
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants Who Experienced Any Dose Limiting Toxicity (DLT)
Description: DLTs were defined as clinically significant adverse events (AEs) (non-hematological, hematological and other events) occurring less than or equal to (<=) 28 days after commencing study treatment and considered to be at least possibly or probably related to study drug by the Investigator. Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (NCI CTCAE v.4.0).
Time Frame: Cycle 1 (Cycle length is 28 days)
Population: Safety analysis set included all participants enrolled and randomized into the Phase 1b of this study, except those who dropped out of the study prior to receiving any study drug, or were without any safety assessment after first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 7
Participants | 1 | 2

2. Primary Outcome: Phase 1b: Cmax: Maximum Observed Plasma Concentration for Golvatinib When Administered in Combination With Sorafenib at Day -7
Time Frame: Day -7: 0-72 hours post-dose
Population: Pharmacokinetic (PK) analysis set was defined as all participants in the safety population who had sufficient concentration data to derive one or more of the PK parameters.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg: Participants received golvatinib 200 mg, tablet, orally, once in combination with sorafenib 400 mg, tablet, orally twice on Day-7.
- Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg: Participants received golvatinib 300 mg, tablet, orally, once in combination with sorafenib 400 mg, tablet, orally twice on Day-7.
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 6
nanograms per milliliter (ng/mL) | 1330 (858) | 2320 (2720)

3. Primary Outcome: Phase 1b: Cmax: Maximum Observed Plasma Concentration for Golvatinib When Administered in Combination With Sorafenib at Day 1 Cycle 1
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length is 28 days)
Population: PK analysis set was defined as all participants in the safety population who had sufficient concentration data to derive one or more of the PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg: Participants received golvatinib 200 mg, tablet, orally, once daily in combination with sorafenib 400 mg, tablet, orally, twice on Day 1 of Cycle 1.
- Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg: Participants received golvatinib 300 mg, tablet, orally, once daily in combination with sorafenib 400 mg, tablet, orally, twice on Day 1 of Cycle 1.
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 6
ng/mL | 1820 (750) | 2820 (3170)

4. Primary Outcome: Phase 1b: Cmax: Maximum Observed Plasma Concentration for Golvatinib When Administered in Combination With Sorafenib at Day 28 Cycle 1
Time Frame: Cycle 1 Day 28: 0-24 hours post-dose
Population: PK analysis set was defined as all participants in the safety population who had sufficient concentration data to derive one or more of the PK parameters. Here, overall number analyzed "N" were the participants who were evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg: Participants received golvatinib 200 mg, tablet, orally, once daily in combination with sorafenib 400 mg, tablet, orally, twice daily from Day 1 to 28 of Cycle 1.
- Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg: Participants received golvatinib 300 mg, tablet, orally, once daily in combination with sorafenib 400 mg, tablet, orally, twice daily from Day 1 to 28 of Cycle 1.
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 4
ng/mL | 2140 (757) | 4570 (3610)

5. Primary Outcome: Phase 1b: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Golvatinib When Administered in Combination With Sorafenib at Day -7
Time Frame: Day -7: 0-72 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 6
hour | 2 [1.03 to 24.3] | 2.38 [1 to 4]

6. Primary Outcome: Phase 1b: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Golvatinib When Administered in Combination With Sorafenib at Day 1 Cycle 1
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length is 28 days)
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 6
hour | 3 [2 to 23.8] | 3.53 [2 to 24]

7. Primary Outcome: Phase 1b: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Golvatinib When Administered in Combination With Sorafenib at Day 28 Cycle 1
Time Frame: Cycle 1 Day 28: 0-24 hours post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 4
hour | 2.98 [1.08 to 4.03] | 5.01 [0.833 to 23.5]

8. Primary Outcome: Phase 1b: AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for Golvatinib When Administered in Combination With Sorafenib at Day -7
Time Frame: Day -7: 0-72 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter(ng*h/mL)
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 6
nanogram*hour per milliliter(ng*h/mL) | 30400 (18900) | 47200 (37500)

9. Primary Outcome: Phase 1b: AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for Golvatinib When Administered in Combination With Sorafenib at Day 1 Cycle 1
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length is 28 days)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 6
ng*h/mL | 24000 (14300) | 36800 (38000)

10. Primary Outcome: Phase 1b: AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for Golvatinib When Administered in Combination With Sorafenib at Day 28 Cycle 1
Time Frame: Cycle 1 Day 28: 0-24 hours post-dose (Cycle length is 28 days)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 4
ng*h/mL | 35300 (16700) | 68700 (72500)

11. Primary Outcome: Phase 1b: t1/2: Terminal Elimination Half-life for Golvatinib When Administered in Combination With Sorafenib at Day -7
Time Frame: Day -7: 0-72 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg
Number analyzed (Participants) | 7 | 6
hour | 38.1 (6.82) | 35.9 (11.7)

12. Primary Outcome: Phase 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to approximately 3 years 11 months)
Population: Safety analysis set included all participants enrolled and randomized to treatment in the Phase 2 of this study, except for those who dropped out prior to receiving any study drug, or were without any safety assessment following the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 42 | 42
Participants
  TEAEs | 42 | 40
  SAEs | 20 | 17

13. Primary Outcome: Phase 2: Number of Participants With AEs by Severity Grades
Description: AE severity was graded using CTCAE version 4.0, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = Severe, Grade 4 = Life-threatening, and Grade 5 = Death related to the AE. All AEs graded as 4 or 5 were considered to be serious. Higher grade indicates more severe condition.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to approximately 3 years 11 months)
Population: Safety analysis set included all participants enrolled and randomized to treatment in the Phase 2 of this study, except for those who dropped out prior to receiving any study drug, or were without any safety assessment following the first dose of study drug. Here, overall number analyzed included are those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 42 | 40
Participants
  Any AE: Grade 1 | 0 | 2
  Any AE: Grade 2 | 4 | 6
  Any AE: Grade 3 | 24 | 25
  Any AE: Grade 4 | 6 | 5
  Any AE: Grade 5 | 8 | 2

14. Primary Outcome: Phase 2: Number of Participants With Adverse Events Related to Vital Signs
Description: Number of participants are reported with AEs related to Vital signs including body temperature, respiratory rate, heart rate, height, and weight.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to approximately 3 years 11 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 42 | 42
Participants | 2 | 0

15. Primary Outcome: Phase 2: Number of Participants With Clinically Significant Change From Baseline in Blood Pressure Including Systolic and Diastolic Blood Pressures
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to approximately 3 years 11 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 42 | 42
Participants | 0 | 0

16. Primary Outcome: Phase 2: Number of Participants With Worst Shifts Post Baseline in Eastern Cooperative Oncology Group Performance Status (ECOG-PS)
Description: Number of participants with worst shifts post baseline in ECOG-PS levels were reported. ECOG has 6 levels (0-5). Level 0 is the best status (fully active, able to carry on all pre-disease performance without restriction); Level 1 is mildly restricted (Restricted in physically strenuous activity but ambulatory ad able to carry out work of a light or sedentary nature, e.g. light house work, office work); Level 2 is more restricted (Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours); Level 3 is restricted (Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours); Level 4 is highly restricted (completely disabled; cannot carry on any selfcare; totally confined to bed or chair); and Level 5 is death (dead).
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to approximately 3 years 11 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 42 | 42
Participants
  ECOG PS Level change from 0 to 1 | 7 | 4
  ECOG PS Level change from 0 to 2 | 3 | 7
  ECOG PS Level change from 0 to 3 | 3 | 0
  ECOG PS Level change from 1 to 2 | 4 | 6
  ECOG PS Level change from 0 to 4 | 0 | 1
  ECOG PS Level change from 1 to 3 | 0 | 5

17. Primary Outcome: Phase 2: Number of Participants With Clinically Significant Change From Baseline in Laboratory Values
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to approximately 3 years 11 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 42 | 42
Participants | 0 | 0

18. Primary Outcome: Phase 2: Number of Participants With Markedly Abnormal Change From Baseline in Electrocardiograms (ECGs) Parameters
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to approximately 3 years 11 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 42 | 42
Participants | 0 | 0

19. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: TTP was defined as the time from the date of randomization until the date of PD of such participants disease based on independent assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. PD was defined as at least a 20% increase or 5 millimeter (mm) increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. TTP was estimated and analyzed using Kaplan-Meier (K-M) method.
Time Frame: From the date of randomization until the date of PD (up to approximately 3 years 11 months)
Population: Modified Intent-to-Treat (MITT) set included all participants randomized in the applicable study arm, except a participant who dropped out of such arm prior to receiving any comparator or investigative drug. Here 'N' (Overall number of participants analyzed) signifies participants with events (PD).
Measure: Median (99% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 31 | 36
weeks | 10.29 [8.57 to 17.14] | 16.00 [8.57 to 23.29]
Statistical Analysis 1: Comparison: Phase 2: Golvatinib 200 mg + Sorafenib 400 mg vs Phase 2: Sorafenib 400 mg; Test type: Superiority; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.56 to 1.50]

20. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization of a participant until (1) the date of first documented progression (2) the date of such participant's death due to any cause based on independent assessments according to RECIST v. 1.1. PD was defined as at least a 20% increase or 5 mm increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. PFS was estimated and analyzed using KM method.
Time Frame: From the date of randomization until the earlier of the following two events: the date of PD or the date of death (Up to approximately 3 years 11 months)
Population: MITT analysis set included all participants randomized in the applicable study arm, except a participant who dropped out of such arm prior to receiving any comparator or investigative drug. Here 'N' (Overall number of participants analyzed) signifies participants with events (PD or/and death).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 32 | 37
weeks | 10.29 [8.14 to 17.14] | 15.57 [8.57 to 23.14]
Statistical Analysis 1: Comparison: Phase 2: Golvatinib 200 mg + Sorafenib 400 mg vs Phase 2: Sorafenib 400 mg; Test type: Superiority; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.57 to 1.50]

21. Secondary Outcome: Phase 2: Percentage of Participants With PFS at Week 12
Description: The PFS rate at week 12 was defined as the percentage of participants who were still alive without disease progression at 12 weeks from the date of randomization. PFS was defined as the time from the date of randomization of a participant until (1) the date of first documented progression (2) the date of such participant's death due to any cause based on independent assessments according to RECIST v. 1.1. PD was defined as at least a 20% increase or 5 mm increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: At 12 weeks
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Groups:
- Phase 2: Golvatinib 200 mg + Sorafenib 400 mg: Participants received golvatinib 200 mg, tablet, orally, once daily in combination with sorafenib 400 mg, tablet, orally, twice daily in 28-days treatment cycles until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 2: Sorafenib 400 mg: Participants received sorafenib 400 mg, tablet, orally, twice daily in 28-days treatment cycles until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 32 | 37
percentage of participants | 47.4 | 57.5

22. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death. Participants were censored at the date of last known alive. OS was analyzed using K-M method.
Time Frame: From the date of randomization until the date of death (Up to approximately 3 years 11 months)
Population: MITT analysis set included all participants randomized in the applicable study arm, except a participant who dropped out of such arm prior to receiving any comparator or investigative drug.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 42 | 42
weeks | 27.86 [20.86 to 67.71] | 37.71 [23.29 to 57.00]
Statistical Analysis 1: Comparison: Phase 2: Golvatinib 200 mg + Sorafenib 400 mg vs Phase 2: Sorafenib 400 mg; Test type: Superiority; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.60 to 1.62]

23. Secondary Outcome: Phase 2: Percentage of Participants With Overall Response
Description: Overall response rate was defined as percentage of participants with best confirmed response (CR) or partial response (PR) assessed by investigator per RECIST v1.1. A confirmatory scan was required after no less than 4 weeks and no later than 8 weeks, starting on the date that the response was first recorded. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<)10 mm. PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization until disease progression or death (Up to approximately 3 years 11 months)
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
Number analyzed (Participants) | 42 | 42
percentage of participant | 4.8 [0.0 to 11.2] | 4.8 [-1.7 to 11.2]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to approximately 3 years 11 months)
Arm/Group | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg | Phase 2: Sorafenib 400 mg
All-Cause Mortality (participants affected / at risk) | 7/7 | 6/7 | 32/42 | 32/42
Serious Adverse Events (participants affected / at risk) | 4/7 | 3/7 | 20/42 | 17/42
Other Adverse Events (participants affected / at risk) | 7/7 | 6/7 | 40/42 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg (N=7) | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg (N=7) | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg (N=42) | Phase 2: Sorafenib 400 mg (N=42)
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Transaminases Increased (Investigations) | 0 | 1 | 0 | 0
Metabolic Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 1 | 0
Nephropathy Toxic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis Psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticular Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Liver Disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Infected Skin Ulcer (Infections and infestations) | 0 | 0 | 1 | 0
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella Infection (Infections and infestations) | 0 | 0 | 0 | 1
Liver Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Scrotal Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 3 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1
Hepatic Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Aneurysm Ruptured (Vascular disorders) | 0 | 0 | 1 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Golvatinib 200 mg + Sorafenib 400 mg (N=7) | Phase 1b: Golvatinib 300 mg + Sorafenib 400 mg (N=7) | Phase 2: Golvatinib 200 mg + Sorafenib 400 mg (N=42) | Phase 2: Sorafenib 400 mg (N=42)
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 26 | 22
Nausea (Gastrointestinal disorders) | 6 | 5 | 15 | 12
Fatigue (General disorders) | 1 | 4 | 13 | 12
Aspartate Aminotransferase Increased (Investigations) | 2 | 5 | 11 | 13
Asthenia (General disorders) | 0 | 1 | 12 | 12
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 | 3 | 15 | 9
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 13 | 9
Vomiting (Gastrointestinal disorders) | 2 | 5 | 14 | 7
Abdominal Pain (Gastrointestinal disorders) | 2 | 5 | 8 | 7
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 4 | 6 | 11
Hypertension (Vascular disorders) | 0 | 1 | 8 | 9
Alanine Aminotransferase Increased (Investigations) | 1 | 4 | 7 | 8
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 8 | 5
Ascites (Gastrointestinal disorders) | 0 | 0 | 8 | 5
Constipation (Gastrointestinal disorders) | 3 | 1 | 7 | 5
Headache (Nervous system disorders) | 0 | 3 | 8 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 9 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 6 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 4 | 5 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 8 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 4 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1
Anaemia Macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 1 | 3 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Anal Fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anorectal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 5 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 6 | 4
Leukopenia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dry Eye (Eye disorders) | 0 | 1 | 2 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 2 | 3 | 5 | 3
Mucosal Inflammation (General disorders) | 1 | 1 | 3 | 3
Pain (General disorders) | 2 | 0 | 0 | 2
Chills (General disorders) | 1 | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0 | 2
Vessel Puncture Site Bruise (General disorders) | 0 | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 2 | 6
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal Candidiasis (Infections and infestations) | 1 | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 3 | 2 | 1 | 2
Blood Bilirubin Increased (Investigations) | 3 | 1 | 3 | 5
Lipase Increased (Investigations) | 1 | 3 | 1 | 7
Ammonia Increased (Investigations) | 0 | 1 | 1 | 1
Amylase Increased (Investigations) | 1 | 0 | 1 | 4
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1 | 1 | 2
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 1 | 0 | 0
Heart Rate Increased (Investigations) | 0 | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 4 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 4 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4 | 3 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 3 | 13 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Fluid Overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 7
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 4 | 3
Hepatic Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 3
Memory Impairment (Nervous system disorders) | 1 | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Restless Legs Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 1 | 2
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 5 | 2
Proteinuria (Renal and urinary disorders) | 2 | 2 | 1 | 2
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal Failure Chronic (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal Polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 4
Lethargy (Nervous system disorders) | 0 | 0 | 3 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Malaise (General disorders) | 0 | 0 | 1 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 2
Transaminases increased (Investigations) | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 2
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Protein urine present (Investigations) | 0 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Acid fast bacilli infection (Infections and infestations) | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric hypomotility (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Genital lesion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Globulins increased (Investigations) | 0 | 0 | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Liver tenderness (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 1
Thyroxine increased (Investigations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vascular insufficiency (Vascular disorders) | 0 | 0 | 1 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Xerosis (General disorders) | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 1 | 3 | 6
Weight Decreased (Investigations) | 0 | 0 | 6 | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 3
Hypotension (Vascular disorders) | 0 | 0 | 2 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 1
Eye Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fungal Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1
Generalised Oedema (General disorders) | 0 | 0 | 0 | 1
Hepatitis C Virus Test Positive (Investigations) | 0 | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Liver Palpable Subcostal (Investigations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes